CLINICAL TRIAL: NCT04035967
Title: Investigation of Parents' Anxiety Level and Health Related Quality of Life in Different Types of Physical Disabilities
Status: Completed | Type: Observational
Sponsor: Sanko University (Other)
Responsible Party: Principal Investigator, Hatice Adıgüzel, Principal Investigator, Sanko University
Other Study IDs: SankoUni
Record Dates: First submitted 2019-07-25; First posted 2019-07-29 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Cerebral Palsy; Down Syndrome; Spina Bifida; Muscular Dystrophy; Parents
Keywords: Physical Disabilities; Anxiety Level; Health Related Quality of Life; Parents'; cerebral palsy
MeSH Terms: conditions — Cerebral Palsy; Down Syndrome; Spinal Dysraphism; Muscular Dystrophies | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Impact on Family Scale (IPFAM), WeeFIM Pediatric Functional Independence Measurement, Nottingham Health Profile. State-Trait Anxiety Inven¬tory (STAI-I and STAI-II), PEDI (Pediatric Evaulation of Disability Inventory)
  Other Names: assesment

SUMMARY:
Disability brings many psychosocial problems in society. The effects of the health of a disabled child on the psychological health and quality of life of the family are inevitable. It has been shown that families with disabled children are exposed to chronic stress, have communication problems and social isolation between parents, and have to spend extra time for the care of children. It is reported in the literature that parents with mentally or physically handicapped children are more stressed and have higher levels of anxiety than parents without children with disabilities. Since activity limitations, participation restrictions, and social and physical barriers are different in each disability group, caregivers may be affected differently. Comparing the quality of life of caregivers of different disability groups and guiding the family in line with the results obtained is important for public health.As the time spent on care may vary in different types of disability, families' levels of distress and anxiety may also be different.There are no studies in the literature comparing the anxiety level of the parents of the individuals with Muscular Dystrophy (MD), Spina Bifida (SB), Cerebral Palsy (SP) and Down Syndrome (DS), which have a very important place in the permanent disability groups, by evaluating the family effect levels and health-related quality of life. . For this reason, this study was planned to investigate the quality of life, anxiety, level of disease and social effects of mothers with different physical disabilities.

DETAILED DESCRIPTION:
Disability is a life-long condition that involves different care needs and includes many psychosocial problems. Having a disabled child is for all family members; creates stress. In the studies, it was found that mothers with disabled children were more stressed and their anxiety levels were higher. There are many disabled people in Turkey and researches related to the caregiver, although there is not enough research on these people. Since activity limitations, participation restrictions and social and physical barriers are different in each disability group, caregivers' influences may also be different. Comparing the quality of life of caregivers of different disability groups and guiding the family in line with the results obtained is important for public health. It is known that the mothers of children with physical disabilities have more symptoms of depression depending on the functional levels of the children. The severity of depression was also found to be higher in people with physical disabilities than other disability groups. In addition, it has been shown that there is a positive relationship between the time spent on care of the child and the level of strain of caregivers. As the time spent on care may vary in different types of disability, families' levels of distress and anxiety may also be different. This is the rehabilitation services; In addition to the physiotherapy applied to physically disabled individuals, it is thought that the social needs of caregivers should be determined and met.In the literature, there are no studies comparing the effects of disease, anxiety levels and quality of life of parents with Muscular Dystrophy (MD), Spina Bifida (SB), Cerebral Palsy (SP) and Down Syndrome (DS). This study was planned to investigate the quality of life, anxiety level, family effects and social effects of the mothers with different physical disabilities.

ELIGIBILITY:
Inclusion Criteria:

* Literate mothers with physical disabilities or healthy children between the ages of 4 and 16, without any known functional and psychological problems
* Literate mothers aged 4-16 years with healthy children, without any known functional and psychological problems
* Signed informed consent form

Exclusion Criteria:

* Mothers of 20 healthy children will be included. with the children who have multiple disabilities
* Mothers of 20 healthy children will be included. with the children who have severe / moderate mental impairment
* Mothers of 20 healthy children will be included. with the children who have Down's syndrome or autism

Ages: 24 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Mothers of 80 cerebral palsy (SP), spina bifida (SP), muscular dystrophy (Duchenne muscular dystrophy (DMD), spinal muscular atrophy (SMA), Becker Muscular Dystrophy (BMD), Down Syndrome will be included.Also mothers of 20 healthy children will be included.
Sampling Method: Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
State-Trait Anxiety Inventory (STAI-I) | first 1 day
  It is a well-researched clinical tool for evaluating the current state of anxiety (State-I).A cut-off point of 39-40 typically indicates clinically significant symptoms of a state of anxiety.
State-Trait Anxiety Inventory (STAI-II). | First 1 day
  STAI-II is a well-researched clinical tool for evaluating the tendency towards anxiety. A cut-off point of 39-40 typically indicates clinically significant symptoms of a state of anxiety.

SECONDARY OUTCOMES:
Nottingham Health Profile | first 1 day
  The NHP is an instrument designed to measure subjective health status containing 38items(answered "yes" or "no") that assess subjective distress in six subgroups:physical mobility (eight items), pain (eight items), sleep (five items), emotional reactions (nine items), social isolation (five items),and energy (three items). Scores for each subgroup range.
  from 0 (no problem) to 100 (all problems listed were present).
Impact on family scale | first 1 day
  The original objective of the Impact on Family Scale is to assess the effect of a child's illness or health condition on the family. All items had astandard four-point scale ranging from strongly agree to strongly disagree.The four factors measured General Negative Impact (11 items), Disruption of Social Relations (nine items), Coping (four items), and Financial Impact (three items).Items are scored on a Likert scale.A low score indicates a higher impact of the chronic disease on the parents. Scores are calculated as percentages according to the highest scores of each part, using inverse proportion computing.
Pediatric Evaluation of Disability Inventory (PEDI) | first 1 day
  PEDI as an evaluative tool capable of detecting the presence, extent, and area of a functional delay in children with physical impairment or combined physical and cognitive impairment. The PEDI comprises three content domains: self-care, mobility, and social function. The self-care domain consists of 73 capability items in 15 skill areas. The mobility domain has 59 items across 13 areas and the social functioning has 65 items across 13 areas. Test items are criterion-referenced; a score of one is achieved if the child is capable of performing the activity in most situations. Higher scores shows better functionality.
The Functional Independence Measure for Children (WeeFIM) | first 1 day
  The WeeFIM was adapted from the adult Functional Independence Measure (FIM), retaining the same structure as the original scale.9 It includes 18 items covering six areas: self-care (eating, grooming, bathing, dressing upper body, dressing lower body, toileting); sphincter control (bladder management, bowel management); transfer (chair ⁄ bed ⁄ wheelchair transfer, toilet transfer, tub ⁄ shower transfer); locomotion (crawling ⁄walking/wheelchair, stair climbing); communication (comprehension, expression); and social cognition (social interaction, problem solving, memory). A 7-level ordinal rating system ranging from 7 (complete independence) to 1 (total assistance), is used to score performance in each item. As with the FIM, the WeeFIM consists of two dimensions: motor and cognitive.The motor scale includes self-care, sphincter control, transfer, and locomotion items; the cognitive scale includes communication, and social cognition items.Higher scores shows better independence.

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Adıgüzel, Principal Investigator — Sanko University; Bülent Elbasan, Ass. Prof., Principal Investigator — Gazi University; Nevin Ergun, Prof., Principal Investigator — Sanko University
Locations (1):
- Sanko University, Gaziantep, Şehitkamil, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No